CLINICAL TRIAL: NCT05054309
Title: A Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Effects of Bifidobacterium Longum NCC3001 on Intestinal and Psychological Symptoms in Subjects With Irritable Bowel Syndrome
Brief Title: A Trial to Evaluate the Effects of Bifidobacterium Longum NCC3001 on Intestinal and Psychological Symptoms in Subjects With Irritable Bowel Syndrome
Acronym: Mood-01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: Syneos Health (Other); Medidata Solutions (Industry); McMaster University (Other); CaligorRx, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 20.01.CLI
Record Dates: First submitted 2021-09-14; First posted 2021-09-23 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: IBS - Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Active Comparator): Bifidobacterium longum [BL NCC3001]
  Interventions: Dietary Supplement: Bifidobacterium longum
- Placebo (Placebo Comparator): Maltodextrin
  Interventions: Dietary Supplement: Bifidobacterium longum

INTERVENTIONS:
Dietary Supplement: Bifidobacterium longum — A Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Effects of Bifidobacterium Longum NCC3001 on Intestinal and Psychological Symptoms in Subjects With Irritable Bowel Syndrome

SUMMARY:
This is a prospective, randomized, placebo-controlled, double-blind, multi-center parallel- design study to evaluate the effect of BL NCC3001 in subjects with Irritable Bowel Syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age between 18 and 70 years inclusive.
2. Willing and able to sign written informed consent prior to study entry.
3. Able to comply with the study procedures, in the opinion of the investigator.
4. Subjects diagnosed with IBS. All subtypes based on Rome IV Criteria with active IBS symptoms as indicated by a score of ≥ 125 on the IBS-SSS.
5. Subjects with psychological symptoms in the absence of a psychiatric diagnosis, defined as a score of 5 to 13 in the depression domain and/or a score of 4 to 9 in the anxiety domain of the DASS-21 questionnaire.

Exclusion Criteria:

1. Concurrent formal diagnosis by a psychiatric specialist, including any mood or anxiety disorder, according to the diagnostic criteria of the Diagnostic and Statistical Manual of Mental Disorders 4th or 5th edition.
2. Concurrent systemic disease and/ or laboratory abnormalities considered by the investigator to be clinically relevant or that could interfere with data collection or interpretation.
3. Concurrent organic gastrointestinal pathology other than benign polyps, diverticulosis, hemorrhoids, lipomas, and melanosis coli.
4. History of attempted suicide in the past 5 years.
5. Previous abdominal surgery except for hernia repair, appendectomy, caesarian section, tubal ligation, hysterectomy, and hemorrhoidectomy.
6. History of substance abuse in the past 2 years, including opiates, phencyclidine, benzodiazepines, amphetamines, cocaine, heroin, alcohol, and cannabinoids (except if medically indicated).
7. Subjects who are on daily treatment with therapeutic doses of drugs having central nervous system effects, including antidepressants and/ or anxiolytics. Low doses of (I) tricyclic antidepressants for abdominal pain/diarrhea related to IBS and (II) anxiolytics used as sleeping pills will be permitted if dose is stable > 3 months prior to the date of randomization.
8. Pregnant or breastfeeding women.
9. Subjects with dementia or other cognitive impairment.
10. Subjects who received antibiotics within the 4 weeks prior to the date of randomization .
11. Known or suspected allergies to the study products.
12. Subjects with increased risk of probiotic sepsis as the following conditions: Immune compromise, including debilitating state or malignancy, central venous catheter, impaired intestinal epithelial barrier (acute diarrheal illness, intestinal inflammation, etc.), cardiac valvular disease.
13. Subjects currently participating or having participated in a therapeutic trial within 3 months prior to the date of randomization.
14. Medically diagnosed lactose intolerance and fructose intolerance without being on a stable lactose or fructose free diet (> 3 months prior to the date of randomization).
15. Medically diagnosed celiac disease.
16. Consumption of any probiotic supplements specified as containing Lactobacillus, Bifidobacteria, Streptococcus, Bacillus coagulans, and Saccharomyces at least 2 weeks prior to the date of randomization.
17. Subjects on regular use of drugs to control IBS symptoms such as bile acid binders (cholestyramine, colestipol or colesevelam, rifaximin, alosetron, lubiprostone, eluxadoline and linaclotide).
18. Recently initiated exclusion diets. Subjects on stable exclusion diets (> 3 months prior to the date of randomization) will not be excluded. This includes subjects with the following diets: gluten-free, lactose-free, paleo, vegetarian, vegan, and low-carbohydrate.
19. Low-FODMAP diet. Subjects on the induction phase of the FODMAP exclusion will not be enrolled. Subjects on the maintenance phase of the diet for more than 3 months prior to the date of randomization with stable diet can be considered for enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2025-02-14 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of Bifidobacterium Longum (BL NCC3001) on Gastrointestinal Symptoms | Baseline to 6 weeks.
  Change from baseline to week 6 in Irritable Bowel Severity Scoring System (IBS-SSS), a questionnaire that includes 5 questions related to the severity of abdominal pain, frequency of abdominal pain, severity of abdominal distention, dissatisfaction with bowel habits, and interference with quality of life over the past 10 days. This cumulative score can therefore range from 0 to 500, with higher scores indicating more severe symptoms.
To evaluate the effect of Bifidobacterium Longum (BL NCC3001) on Psychological Symptoms | Baseline to 6 weeks.
  Change from baseline to week 6 in Hospital Anxiety and Depression Scale (HADS-Total) score, a 14-item scale assessing two dimensions (anxiety and depression, 7 items for each) of psychological distress. Each item is scored from 0-3 in a Likert manner. Outcome measures are the anxiety score (0-21), depression score (0-21) and the total score (0-42).

SECONDARY OUTCOMES:
Hospital Anxiety Depression Scale - Depression (HADS-D) score | Day -1, Day 43 (± 2 days)
  Change from baseline to Week 6 in Hospital Anxiety Depression Scale-Depression (HADS-D) score, a 14-item scale assessing depression (7 items) of psychological distress. Each item is scored from 0-3 in a Likert manner. Outcome measures are the depression score (0-21).
Hospital Anxiety Depression Scale - Anxiety (HADS-A) score | Day -1, Day 43 (± 2 days)
  Change from baseline to Week 6 in Hospital Anxiety Depression Scale-Anxiety (HADS-A) score, a 14-item scale assessing anxiety (7 items) of psychological distress. Each item is scored from 0-3 in a Likert manner. Outcome measures are the anxiety score (0-21).
Depression Anxiety Stress Scale (DASS-21) | Day -1, Day 43 (± 2 days)
  Change from baseline to Week 6 in Depression Anxiety Stress Scale (DASS-21), a four-point Likert scale ranging from 0 ("did not apply to me at all") to 3 ("applied to me very much" or "most of the time"). The outcome measures correspond to the total scores (0-21) of the subscales.
Perceived Stress Scale (PSS) | Day -1, Day 43 (± 2 days)
  Change from baseline to Week 6 in Perceived Stress Scale (PSS), includes several direct queries about current levels of experienced stress, each item is rated on a Likert scale (0-4), the range of the total score is 0-40.
Irritable Bowel Severity Scoring System (IBS-SSS) Pain severity | Day -1, Day 43 (± 2 days)
  Change from baseline to Week 6 in Irritable Bowel Severity Scoring System (IBS-SSS) pain severity, a question related to the severity of abdominal pain over the past 10 days. The question is scored on a 100-point visual analogue scale, which is anchored with the 2 extremes (e.g., no pain on the far left to severe pain on the far right).
Irritable Bowel Severity Scoring System (IBS-SSS) Pain frequency | Day -1, Day 43 (± 2 days)
  Change from baseline to Week 6 in Irritable Bowel Severity Scoring System (IBS-SSS) pain frequency, a question related to the frequency of abdominal pain over the past 10 days. The question is scored on a 100-point visual analogue scale, which is anchored with the 2 extremes (e.g., no pain on the far left to severe pain on the far right).
Irritable Bowel Severity Scoring System (IBS-SSS) Bloating severity | Day -1, Day 43 (± 2 days)
  Change from baseline to Week 6 in Irritable Bowel Severity Scoring System (IBS-SSS) bloating severity, a question related to the severity of abdominal distention over the past 10 days. The question is scored on a 100-point visual analogue scale, which is anchored with the 2 extremes (e.g., no pain on the far left to severe pain on the far right).
Irritable Bowel Severity Scoring System (IBS-SSS) Bowel habit | Day -1, Day 43 (± 2 days)
  Change from baseline to Week 6 in Irritable Bowel Severity Scoring System (IBS-SSS) bowel habit, a question related to dissatisfaction with bowel habits over the past 10 days. The question is scored on a 100-point visual analogue scale, which is anchored with the 2 extremes (e.g., no pain on the far left to severe pain on the far right).
Irritable Bowel Severity Scoring System (IBS-SSS) Life impact | Day -1, Day 43 (± 2 days)
  Change from baseline to Week 6 in Irritable Bowel Severity Scoring System (IBS-SSS) life impact, a question related to interference with quality of life over the past 10 days. The question is scored on a 100-point visual analogue scale, which is anchored with the 2 extremes (e.g., no pain on the far left to severe pain on the far right).
Irritable Bowel Syndrome Quality of Life questionnaire (IBS-QoL) | Day -1, Day 43 (± 2 days)
  Change from baseline to Week 6 in Irritable Bowel Syndrome Quality of Life questionnaire (IBS-QoL), a 34-item, validated, condition-specific measure based on 5-point Likert scale for assessing health-related quality of life in the past month among persons with IBS.
Patient Health Questionnaire (PHQ-12) | Day -1, Day 43 (± 2 days)
  Change from baseline to Week 6 in Patient Health Questionnaire (PHQ-12), each somatic symptom is evaluated in a Likert scale from 0 to 2 (not bothered at all, bothered a little and bothered a lot) giving a maximum total of 24 points.
Sheehan Disability Scale (SDS) | Day -1, Day 43 (± 2 days)
  Change from baseline to Week 6 in Sheehan Disability Scale (SDS), the patients rates the extent to which work/school, social and family life are impaired by his/her symptoms on a 10-point VAS.
Amount of Bifidobacterium Longum (BL NCC3001) present in stool | Day -1, Day 43 (± 2 days)
  Change from baseline to Week 6
Irritable Bowel Severity Scoring System (IBS-SSS) score | Day -1, Day 71 (± 2 days)
  Change from baseline to Week 10 in Irritable Bowel Severity Scoring System (IBS-SSS) score, a cumulative score which can therefore range from 0 to 500, with higher scores indicating more severe symptoms. Mild, moderate, and severe cases are indicated by scores of 75 to 175.
Hospital Anxiety Depression Scale (HADS) total score | Day -1, Day 71 (± 2 days)
  Change from baseline to Week 10 in Hospital Anxiety Depression Scale (HADS) total score, a 14-item scale assessing two dimensions (anxiety and depression, 7 items for each) of psychological distress. Each item is scored from 0-3 in a Likert manner. Outcome measures are the anxiety score (0-21), depression score (0-21) and the total score (0-42).
Rescue Medication | Day 43 (± 2 days)
  Difference in proportions compared to placebo at Week 6
Psychological distress improvement according to the Patient's Global Impression of Change of "Psychological Distress" | Day 43 (± 2 days)
  Difference in proportions compared to placebo at Week 6 using a 7-point Likert scale depicting a patient's rating of overall improvement of the psychological distress since the beginning of treatment. The range of the score is 1 to 7.
Active treatment randomization perception: "Do you think you have taken the placebo or active treatment?" | Day 43 (± 2 days)
  Difference in proportions compared to placebo at Week 6

OTHER OUTCOMES:
Microbiota composition - A subset of 80 subjects (40 per arm) | Day -1, Day 43 (± 2 days), Day 71 (± 2 days)
  Changes in microbiota composition in feces
Microbiota metabolic activity in feces - A subset of 80 subjects (40 per arm) | Day -1, Day 43 (± 2 days)
  Changes in microbiota metabolic activity in feces
Microbiota metabolic activity in blood - A subset of 80 subjects (40 per arm) | Day -1, Day 43 (± 2 days)
  Changes in microbiota metabolic activity in blood
Microbiota metabolic activity in urine - A subset of 80 subjects (40 per arm) | Day -1, Day 43 (± 2 days)
  Changes in microbiota metabolic activity in urine
Cortisol levels in saliva - A subset of 80 subjects (40 per arm) | Day -1, Day 43 (± 2 days)
  Change in cortisol levels in saliva
Biomarkers in blood - A subset of 80 subjects (40 per arm) | Day -1, Day 43 (± 2 days)
  Detection of Biomarkers in blood
Neurotransmitters in blood - A subset of 80 subjects (40 per arm) | Day -1, Day 43 (± 2 days)
  Detection of Neurotransmitters in blood
Amount of Bifidobacterium Longum (BL NCC3001) in stool | Day 71 (± 2 days)
  Amount of Bifidobacterium Longum (BL NCC3001) in stool

CONTACTS AND LOCATIONS:
Overall Officials: Premsyl Bercik, MD, Principal Investigator — McMaster University
Locations (11):
- Canada (11):
  - University of Calgary, Calgary, Alberta
  - University Of Alberta, Edmonton, Alberta
  - Eastern Regional Health Authority, St. John's, Newfoundland and Labrador
  - Medicor Research Inc., Greater Sudbury, Ontario
  - McMaster University, Hamilton, Ontario
  - Scott Shulman Medicine Professional Corporation, North Bay, Ontario
  - The Ottawa Hospital General Campus, Ottawa, Ontario
  - Canadian Phase Onward Inc., Toronto, Ontario
  - Diex Recherche Quebec Inc., Québec, Quebec
  - DIEX Recherche, Saint-Charles-Borromée, Quebec
  - PerCuro Clinical Research Ltd., Victoria

IPD SHARING:
Plan to Share IPD: No